CLINICAL TRIAL: NCT02682550
Title: Analysis of the Danger Response After Polytrauma Based on the National Polytrauma-serum-bank of the Trauma Research Network (NTF) of the German Society for Orthopaedics and Trauma (DGOU)
Brief Title: Danger Response in Polytrauma Patients
Acronym: NTF-PT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Markus Huber-Lang, M.D., Professor for Clinical and Experimental Trauma-Immunology, University of Ulm
Other Study IDs: NTF_PT_2014
Record Dates: First submitted 2016-01-19; First posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Trauma
Keywords: polytrauma; hemorrhagic shock; sepsis; MODS
MeSH Terms: conditions — Multiple Trauma; Shock, Hemorrhagic; Sepsis; Multiple Organ Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA-Plasma and Serum (drawn from polytrauma patients with an injury severity score ≥25)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ctrl: healthy volunteers, sex- and age matched Blood drawing at one time point: 20 ml
  Interventions: Procedure: blood drawing
- PT: polytrauma patients fulfilling the following criteria:
  * injury severity score ≥25
  * age ≥ 18 Blood drawing at admission to the emergency room, 8 h, 24h, 48 h, 120 h and 240 h post trauma: 20 ml
  Interventions: Procedure: blood drawing

INTERVENTIONS:
Procedure: blood drawing — blood drawing

SUMMARY:
The NTF_PT_2014 multicenter study aims to collect, store, and analyse plasma and serum from polytrauma-patients (injury severity score ≥25) and corresponding clinical data to address 1) how trauma modulates the release of danger molecules, inflammatory mediators, coagulation factors and novel biomarkers, 2) how the specific injury pattern affects the posttraumatic response and regenerative potential on an organ-, cell, and molecular level, and 3) how could a specific organ- and immune-monitoring predict the clinical outcome.

DETAILED DESCRIPTION:
Polytrauma is worldwide a major socio-economic problem. Especially the polytrauma-induced complications, such as systemic inflammatory response, sepsis, organ dysfunction remain associated with a high morbidity and mortality rate. The underlying posttraumatic pathophysiology remains poorly understood, especially since the polytrauma patients present a highly variable patient cohort with complex injury patterns, comorbidities and different therapeutic strategies.

Therefore, the present "NTF_PT_2014" multicenter study of the Trauma Research Network (NTF) of the German Society for Orthopaedics and Trauma (DGOU) with its established national Polytrauma-serum-bank aims to collect, store, and analyse plasma and serum from polytrauma-patients and corresponding clinical data to address:

1. how trauma modulates the release of danger molecules, inflammatory mediators, coagulation factors and novel biomarkers?
2. how the specific injury pattern affects the posttraumatic response and regenerative potential on a organ-, cell, and molecular level?
3. how could a specific organ- and immune-monitoring predict the clinical outcome?

Blood will be drawn from anticipated 1000 patients with an injury severity score ≥ 25 at the time of hospital admission (in the emergency room), 8 h, 24h, 48, 120 h, and 240 h post injury. The biochemical and immune-monitoring data will be correlated to corresponding clinical data and data from the German Trauma Registry (TraumaRegister DGU®).

Blood from age- and sex matched healthy volunteers (n=200) will serve as a control group.

The study will provide a detailed picture of the molecular danger response after multiple injury and may reveal novel therapeutic targets for posttraumatic complications.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* healthy

Exclusion Criteria:

* age < 18
* gravidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: polytrauma patients age ≥ 18 ISS ≥ 25
  Exclusion: cardiopulmonary reanimation before admission, gravidity, no chemotherapy or radiotherapy within the last 3 months, immune supressive drugs, hemodialysis, age < 18
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) plasma concentration | 24 hours after polytrauma
  Interleukin-6 may indicate the extent of tissue damage and the inflammatory response after trauma

SECONDARY OUTCOMES:
Multiple-Organ-Failure (MOF) | 0-28 days after trauma
  daily "Sequential Organ Failure Assessment" score
Sepsis | 0-28 days after trauma
  sepsis definition daily in accordance to the "American College of Chest Physicians/Society of Critical Care Medicine" Consensus
S100 calcium-binding protein B plasma concentration | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  plasma S100 calcium-binding protein B as a marker for central nervous system injury
Creatinine plasma concentration | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  plasma creatinine to measure the glomerular filtration rate as a marker of renal function.
Bilirubin plasma concentration | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  plasma bilirubin as a biomarker for liver failure
Survival | 28-day survival
  survival recorded every day: yes/no
monomeric C-reactive protein | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  C-reactive protein may not only represent a biomarker of the systemic inflammatory response after trauma but also help to clear danger- and pathogen-associated molecular patterns
pentameric C-reactive protein | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  C-reactive protein may not only represent a biomarker of the systemic inflammatory response after trauma but also help to clear danger- and pathogen-associated molecular patterns
Interleukin-10 | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  Inflammatory profiling: plasma concentrations of Interleukin-10
Interleukin-1beta | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  Inflammatory profiling: plasma concentrations of Interleukin-1beta
Complement factor C3a | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  Inflammatory profiling: plasma concentrations of Complement factor C3a
Arterial partial oxygen pressure | daily, the first 10 days after trauma
  Arterial partial oxygen pressure reflects lung performance
Number of microvesicles derived from granulocytes in plasma of patients (as assessed by flow cytometry) | within 30 minutes after polytrauma/ 8 hours/ 24 hours/ 48 hours/ 120 hours/240 hours after polytrauma
  Microvesicles as carriers of clotting factors and inflammatory molecules may be significantly involved in the coagulatory and inflammatory response after trauma

CONTACTS AND LOCATIONS:
Overall Officials: Markus Huber-Lang, M.D. Prof, Study Director — University of Ulm, Center for Biomedical Research (ZBF)
Locations (1):
- University Hospital, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halbgebauer R, Karasu E, Braun CK, Palmer A, Braumuller S, Schultze A, Schafer F, Buckle S, Eigner A, Wachter U, Radermacher P, Resuello RRG, Tuplano JV, Nilsson Ekdahl K, Nilsson B, Armacki M, Kleger A, Seufferlein T, Kalbitz M, Gebhard F, Lambris JD, van Griensven M, Huber-Lang M. Thirty-Eight-Negative Kinase 1 Is a Mediator of Acute Kidney Injury in Experimental and Clinical Traumatic Hemorrhagic Shock. Front Immunol. 2020 Aug 26;11:2081. doi: 10.3389/fimmu.2020.02081. eCollection 2020. PMID 32983160